CLINICAL TRIAL: NCT03970603
Title: Weight-Bearing Timing and Outcomes After Surgical Suture Button Repair of the Distal Tibiofibular Syndesmosis
Brief Title: Syndesmosis Ankle Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyle Schweser MD (Other)
Responsible Party: Sponsor-Investigator, Kyle Schweser MD, Orthopaedic Trauma Surgeon, Assistant Professor, University of Missouri-Columbia
Organization: University of Missouri-Columbia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014428
Record Dates: First submitted 2019-05-28; First posted 2019-05-31 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Syndesmotic Disruption; Weight-bearing Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Weight-Bearing (Active Comparator): Being directed to bear weight on the affected ankle two weeks from suture button fixation for syndesmotic disruption
  Interventions: Other: Early Weight-Bearing
- Delayed/Late Weight-Bearing (Active Comparator): Being directed to bear weight on the affected ankle six weeks from suture button fixation for syndesmotic disruption
  Interventions: Other: Delayed/Late Weight-Bearing

INTERVENTIONS:
Other: Early Weight-Bearing — Being directed to bear weight on the affected ankle two weeks from suture button fixation for syndesmotic disruption
  Arms: Early Weight-Bearing
Other: Delayed/Late Weight-Bearing — Being directed to bear weight on the affected ankle six weeks from suture button fixation for syndesmotic disruption
  Arms: Delayed/Late Weight-Bearing

SUMMARY:
A debate regarding ankle fracture fixation centers on time to weight bearing. Recent literature has supported immediate weight bearing in surgically stabilized ankle fractures. However, significant variation among orthopaedic surgeons persists, and weight bearing recommendations change when there is a syndesmotic disruption. There is very little literature on time to weight bearing, with most available series casting/immobilizing these injuries for 6 weeks after fixation. There is very little data examining post-operative weight bearing after syndesmotic stabilization, and the majority centers on screw fixation. The minimum time to weight bearing after an ankle fracture with syndesmotic fixation in the literature is 4 weeks, with most focusing on 6 to 12 weeks. Based on biomechanical data regarding suture button techniques, the investigators hypothesize that patients undergoing ankle fracture fixation plus suture button fixation of their syndesmotic disruption will be able to safely bear weight early (2 weeks) after surgery. The investigator's null hypothesis is that there will be no difference between early weight bearing (2 weeks), and late weight bearing (6 weeks) in terms of outcome, hardware failure, loss of reduction, and return to work.

Adult patients who have an ankle fracture with suspected syndesmotic disruption, requiring a suture button fixation operative intervention will be randomized into early (2 weeks post-surgically) weight-bearing status or delayed weight-bearing status (non-weight-bearing for 6 weeks following fixation).

Primary objective: Maintenance of ankle reduction at 1 year follow-up (measured by comparing immediate post-op CT and 1 year time-point CT).

Secondary Objectives: Pain scores, surgical experience, work productivity and activity impairment , AAOS foot and ankle scores (2w, 6w, 12w, 6m, 1y), use of assistive devices, range of motion, physical therapy requirement/length of use/compliance, post-operative protocol compliance, post-operative complications (wound healing, infection, implant failure, fracture healing).

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Ankle fracture with suspected syndesmotic disruption that would likely be treated with suture button fixation operative intervention
3. Ability to ambulate preoperatively

Exclusion Criteria:

1. Younger than 18
2. Length unstable syndesmotic injury (i.e. Maisonneuve)
3. Neuropathic diabetics
4. 325 pounds or more
5. Prisoner
6. Pregnant or lactating
7. End stage renal disease
8. Inability to follow commands (dementia, TBI, etc.)
9. Polytrauma patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2023-10-26 (Actual); Study Completion 2025-09-25 (Actual)

PRIMARY OUTCOMES:
Measure of the syndesmotic change | 1 year
  Determined by comparing the 1-year, post-operative CT scan to the immediate post-operative CT scan of the injured ankle

SECONDARY OUTCOMES:
Pain scores | 2 weeks to 1 year
  Measured on a 0-10 scale by VAS or PROMIS patient reported outcome forms
Surgical Experience (SSQ-8) | Day 0
  The SSQ-8 (Surgical Satisfaction Score) is a patient administered 8-item survey designed to asses satisfaction after a surgical procedure. Answers are then measured on a scale of 1 to 5 or 6, with 1 being the best outcome score.
Work productivity and activity impairment (WPAI) | 6 weeks to 1 year
  The Work Productivity and Activity Impairment (WPAI) questionnaire is a self-administered instrument used to assess the impact of disease on productivity. The sum of specific health problem impairment and impairment due to other health reasons is equal to impairment due to all health reasons. WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity, i.e., worse outcomes.
Foot and ankle outcomes (AAOS) | 2 weeks to 1 year
  The AAOS foot and ankle questionnaire is a patient-administrated 25-item survey specifically developed for foot and ankle-related disability. The questionnaire is divided into two scales, the Foot and Ankle Core scale, comprised of 20 questions and the Shoe Comfort Scale with five questions. The questions themselves are distributed amongst five different categories: Pain (9 items), function (6 items), stiffness and swelling (2 items), giving way (3 items) and shoe comfort (5 items). Answers are then measured on a scale of 1 to 5 or 6, with1 being the best outcome score.

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Schweser, MD, Principal Investigator — University of Missouri Health System, Department of Orthopaedic Surgery
Locations (1):
- Vicki Jones, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided